CLINICAL TRIAL: NCT02150226
Title: Low Thermal Degradation of Monolithic Zirconia Prostheses: an up to 5-year Original Prospective Clinical Study Using ex Vivo Analyses
Brief Title: Y-TZP and In-mouth Low Thermal Degradation: A Prospective Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Liege (Other)
Collaborators: DMG Paris Descartes (Other)
Responsible Party: Principal Investigator, Mainjot Amélie, Doctor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FZ001
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Zirconia Monolithic Dental Restorations: In-mouth Behaviour, LTD and Wear
MeSH Terms: interventions — Crowns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: Zirconia monolithic crowns and bridges (Experimental): Evaluation of Lava Plus zirconia dental crowns and bridges
  Interventions: Device: Lava plus (3M) crowns and bridges

INTERVENTIONS:
Device: Lava plus (3M) crowns and bridges — Zirconia monolithic dental crowns and bridges evaluation

SUMMARY:
The objective of this work is to study in-mouth aging and LTD of monolithic zirconia restorations. Microstructural changes characteristic of LTD processes, wear, and clinical behaviour following standard parameters will be evaluated. Notably Raman spectroscopy and 3D laser surface analysis will be used, directly on the restorations, which will be removed at regular intervals.The working hypothesis is that LTD process is very slow at the scale at the lifespan of dental prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Full zirconia crowns in the posterior region (molar/premolar)
* On teeth or implants
* Single unit restorations cemented on natural teeth and implants (including screw-retained restorations if possible, but no internal connections)
* Multi-unit restorations on implants
* If nightguard: to be performed on the antagonist

Exclusion Criteria:

* Patients with removable prosthesis as an antagonist

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
in-mouth LTD of monolithic zirconia restorations on natural teeth and implants | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Dentistry University of Liege, Liège, Belgium

REFERENCES:
- [Derived] Koenig V, Douillard T, Chevalier J, Amiard F, Lamy de la Chapelle M, Le Goff S, Vanheusden A, Dardenne N, Wulfman C, Mainjot A. Intraoral low-temperature degradation of monolithic zirconia dental prostheses: 5-year results of a prospective clinical study with ex vivo monitoring. Dent Mater. 2024 Feb;40(2):198-209. doi: 10.1016/j.dental.2023.11.008. Epub 2023 Nov 10. PMID 37951752
- [Derived] Koenig V, Wulfman CP, Derbanne MA, Dupont NM, Le Goff SO, Tang ML, Seidel L, Dewael TY, Vanheusden AJ, Mainjot AK. Aging of monolithic zirconia dental prostheses: Protocol for a 5-year prospective clinical study using ex vivo analyses. Contemp Clin Trials Commun. 2016 Jun 17;4:25-32. doi: 10.1016/j.conctc.2016.06.001. eCollection 2016 Dec 15. PMID 29736467